CLINICAL TRIAL: NCT01843101
Title: Investigation of Different Scanning Protocols for 3 Dimensional High-resolution Imaging of the Human Cornea With Optical Coherence Tomography (OCT) - A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-040413
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Corneal Neovascularisation; Keratoconus
Keywords: Optical Coherence Tomography; Cornea; Imaging
MeSH Terms: conditions — Corneal Neovascularization; Keratoconus; Corneal Diseases | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy volunteers (Other): 10 healthy volunteers
  Interventions: Device: Optical Coherence Tomography
- Corneal Neovascularisation (Other): 5 patients with corneal neovascularisation
  Interventions: Device: Optical Coherence Tomography
- Keratoconus (Other): 5 patients with keratoconus
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Imaging of the cornea using ultrahigh resolution Spectral Domain OCT

SUMMARY:
The aim of the present study is to develop a protocol for optimal corneal 3-dimensional imaging based on measurements in healthy volunteers. For this purpose, a customized ultra-high resolution Spectral Domain OCT will be used. To validate whether the protocol can also be applied in patients with corneal pathologies, for whom it is intended to be used, measurements in these patients will be performed. We propose to obtain images from patients with keratoconus, since this is one of the most frequent causes for corneal transplantations in Europe and from patients with corneal neovascularization which is a major cause of vision loss in several ophthalmic diseases. Based on the obtained measurement protocol, further studies investigating the pathophysiology or treatment success of several corneal pathologies can be planned.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Men and women aged over 18 years
* Normal findings in the slit lamp examination, no corneal pathologies

Patients with keratoconus:

* Men and women aged over 18 years
* Presence of keratoconus
* No ophthalmic surgery in the 3 months preceding the study

Patients with corneal neovascularization:

* Men and women aged over 18 years
* Presence of corneal neovascularization
* No ophthalmic surgery in the 3 months preceding the study

Exclusion Criteria:

* Participation in a clinical trial in the previous 3 weeks
* Presence of any abnormalities preventing reliable measurements as judged by the investigator
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Corneal Imaging | 1 day
  Development of a measurement protocol for 3 dimensional imaging of the human cornea

SECONDARY OUTCOMES:
Imaging of corneal pathologies | 1 day
  Application of the protocol in patients with corneal pathologies

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Napora, MD, PhD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria